CLINICAL TRIAL: NCT01397227
Title: A Phase I/IIa, Double-blind, Randomized, Placebo-controlled, Dose-escalation Clinical Study Evaluating Safety, Tolerability and Immunogenicity of Two Dose Levels of Recombinant Adenoviral Serotype Ad35 and Serotype Ad26 Vectors Expressing the Malaria Plasmodium Falciparum Circumsporozoite Antigen Administered as Heterologous Prime-boost Regimen, and Assessing Protective Efficacy of the Higher Dose in a Malaria Challenge Model in Unblinded Conditions
Brief Title: A Study to Assess the Immunogenicity, Tolerability and Safety of a Malaria Vaccine and Also Its Protective Efficacy in a Malaria Challenge Model
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MAL-V-A001
Record Dates: First submitted 2011-07-12; First posted 2011-07-19 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-09

CONDITIONS: Malaria
Keywords: Malaria; Plasmodium falciparum; Vaccination; Prophylaxis; Adenovirus
MeSH Terms: conditions — Malaria; Malaria, Falciparum; Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (Low Dose) (Experimental): Ad35.CS.01/Ad26.CS.01 - 1 x 10^10 vp
  Interventions: Biological: Ad35.CS.01/Ad26.CS.01 low dose (1 x 10^10 vp)
- Cohort 2 (High Dose) (Experimental): Ad35.CS.01/Ad26.CS.01 - 5 x 10^10 vp
  Interventions: Biological: Ad 35.CS.01/Ad 26.CS.01 high dose (5 x 10^10 vp)
- Cohort 1 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- Cohort 2 - Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad35.CS.01/Ad26.CS.01 low dose (1 x 10^10 vp) — Prime-boost schedule: Each subject receives two injections of Ad35.CS.01 (on Days 0 and 28) followed by one injection of Ad26.CS.01 (on either Day 55 or 59).
  Arms: Cohort 1 (Low Dose)
Biological: Ad 35.CS.01/Ad 26.CS.01 high dose (5 x 10^10 vp) — Prime-boost schedule: Each subject receives two injections of Ad35.CS.01 (on Days 0 and 28) followed by one injection of Ad26.CS.01 (on either Day 55 or 59).
  Arms: Cohort 2 (High Dose)
Biological: Placebo — Each placebo subject receives in total three injections of placebo: Day 0, Day 28, and either Day 55 or 59
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of two dose levels (1x10^10 and 5x10^10 virus particles (vp)) of the adenovirus serotype (Ad) Ad35.CS.01/Ad26.CS.01 prime-boost malaria candidate vaccine, followed by an evaluation of the protective efficacy of the higher dose level in an experimental malaria challenge.

The study will be in 3 phases:

1. a dose escalation / vaccination phase in which both dose levels will be tested
2. a malaria challenge phase in which only subjects receiving the Ad35.CS.01/Ad26.CS.01 5x10^10 vp dose level, together with six infectivity control subjects, will be exposed to experimental challenge with Plasmodium falciparum
3. a long term follow up phase in which all subjects who received active vaccine from both dose levels and/or malaria challenge will be included

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects aged ≥18 to ≤50 years on Study Day 0.
* Able and willing to participate for the duration of the study, to comply with protocol provisions and to undergo malaria challenge.
* Able and willing to provide written informed consent.
* Free of obvious health-problems as established by medical history, physical examination, laboratory assessment and clinical judgment of the investigator.
* If the participant is biologically female she must:

  * Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test performed at screening within 7 days before the 1st vaccine administration, and agree to a urine β-hCG pregnancy test at Study Day 0 and at each subsequent vaccine administration, before the challenge period, and at the end of the challenge period.
  * Agree to consistently use effective contraception from 21 days prior to Study Day 0 for the duration of the study, for sexual activity that could lead to pregnancy.
  * Agree to not seek pregnancy through alternative methods such as artificial insemination or in vitro fertilization until after the last scheduled protocol visit.
* Male subjects engaged in sexual activities which could lead to pregnancy must agree to use a reliable barrier contraceptive plus spermicide for the duration of the study.

Exclusion Criteria:

* Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have implications for current health status in the opinion of the Investigator. A clinically significant condition or process includes but is not limited to:
* A process that would affect the immune response,
* A process that would require medication that affects the immune response,
* Any contraindication to repeated phlebotomy,
* A condition or process in which signs or symptoms could be confused with reactions to vaccination or malaria challenge and/or infection, including dermatologic abnormalities at the site of sporozoite inoculation/vaccination, or
* Any condition specifically listed among the exclusion criteria below.
* Clinically significant acute illness, including oral temperature >38.0 °C, or infection within 2 weeks of Study Day 0 that, in the opinion of the Investigator, would interfere with study assessments or cause significant implications for subject safety.
* History of, or known active cardiac disease including: (1) prior myocardial infarction (heart attack); (2) angina pectoris; (3) congestive heart failure; (4) valvular heart disease; (5) cardiomyopathy; (6) pericarditis; (7) stroke or transient ischemic attack; (8) exertional chest pain or shortness of breath; or (9) other heart conditions under the care of a doctor.
* Elevated (moderate or high) risk of coronary heart disease as determined by the NHANES I cardiovascular risk assessment criteria.
* Clinically significant ECG findings, as determined by the study cardiologist.
* History of malignancy, including hematologic and skin cancers (except for a localized basal cell carcinoma).
* History of coagulation defects or bleeding that can not be linked to trauma or surgery.
* History of receiving blood or blood products (such as blood transfusions, platelet transfusion, immunoglobulins, hyperimmune serum) within 6 months prior to Study Day 0.
* History of mental illness as defined by symptoms interfering with social or occupational function or suicidal thoughts / attempts, excluding minor depression resolved or successfully treated at least 3 years prior to Study Day 0.
* Any clinically significant history of known or suspected anaphylaxis or hypersensitivity reaction to vaccinations.
* History of splenectomy.
* Clinically significant screening laboratory abnormalities within 90 days of Study Day 0.
* Positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg).
* Positive Neutralizing Antibody titers (IC90 >16) against Ad26 and/or Ad35.
* Pregnant or lactating female.
* Chronic (longer than 14 days) administration of immunosuppressants (including oral or inhaled) or other immune-modifying drugs within 6 months prior to Study Day 0, including oral corticosteroids in dosages of ≥0.5 mg/kg/day prednisone or equivalent.
* Blood donation (typical US blood volume donations are 470 mL) or significant blood loss (defined as total cumulative volume >500 mL, including screening blood volumes) within 56 days before first dosing or plasma donation within 7 days prior to Study Day 0.
* Vaccination with a live vaccine within 30 days prior to Study Day 0 or with a non-replicating, inactivated or subunit vaccine within 14 days prior to Study Day 0 or planned vaccination of any type during the study period.
* Prior receipt of a malaria vaccine.
* Any history of malaria diagnosed on positive blood smear.
* Use of antimalarial prophylaxis, or travel to a malaria endemic region within 6 months prior to Study Day 0.
* Any history of residence (>3 months) in area known to have significant transmission of Plasmodium falciparum.
* Planned travel to a malaria endemic region during the study period.
* Prior receipt of a recombinant adenovirus vector vaccine.
* Known hypersensitivity to components of the vaccine or proposed antimalarial medications.
* Employee at the malaria clinical trial center or investigator or relative children or spouse of any investigator.
* Identification of any condition or finding that, in the opinion of the investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of study endpoints or would jeopardize the rights, safety or welfare of the subject participating in the study.
* Smokers with current use of >10 cigarettes/day or >15 pack-years of lifetime cigarette use.
* Known history of hemoglobinopathy.
* Suspected or known alcohol or drug abuse as defined by the American Psychiatric Association in the DSM IV.
* Ocular disease defined as retinopathy or visual field defects.
* Chronic neurological symptoms including seizures or migraine headaches.
* Concurrent participation in other investigational protocols or in receipt of an investigational product within the previous 6 months of Study Day 0 or planned receipt of another investigational product during the course of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Solicited local and systemic adverse events (AEs) | For 7 days after each vaccination and at each visit during the challenge period
  Type and frequency of solicited local and systemic AEs to be recorded. Solicited AEs in the challenge period are collected via a reactogenicity checklist during study visits. Solicited AEs in the vaccination period are collected via a Subject Diary.
Unsolicited AEs | At each visit during the vaccination period
  Type and frequency of unsolicited AEs to be recorded
Vital signs | Before and after each vaccination during the vaccination period, before and after malaria challenge and at each visit during the challenge period
  Temperature (oral), pulse, respiratory rate, blood pressure and pulse oximetry will be measured
Changes in laboratory parameters from baseline to end of vaccination phase | Screening/baseline, 7 days after each vaccination, and Days 101 and 115 of the challenge period
  Assessment made on the changes in each laboratory parameter from baseline to the end of the vaccination phase at each time point. Parameters measured:
  Biochemistry: glucose, potassium, creatinine, γ-glutamyl transferase, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, C-reactive protein and erythrocyte sedimentation rate.
  Hematology: hemoglobin, hematocrit, white blood cell count, white blood cell differential, red blood cell count and platelet count.
  Urinalysis: leucocytes, blood, protein, ketones and glucose (by dipstick).

SECONDARY OUTCOMES:
Immunogenicity | Blood samples drawn at baseline (screening) and Study Days 14, 28, 42, 55/59, 69/73, 86 and 115
  * Anti-circumsporozoite antibodies will be assessed by enzyme-linked immunosorbent assay
  * T-cell responses against circumsporozoite protein will be assessed by ELISPOT assays and flow cytometry
  * Neutralizing antibodies to Ad26, and Ad35 will be assessed by neutralizing antibody assay
Efficacy - patent parasitemia | Vaccine recipients are monitored for the development of parasitemia for 28 days post-malaria challenge
  Development of patent parasitemia diagnosed on peripheral blood smear

CONTACTS AND LOCATIONS:
Overall Officials: Angela Talley, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Malaria Clinical Trials Center at Seattle Biomedical Research Institute, Seattle, Washington, United States